CLINICAL TRIAL: NCT02635009
Title: Randomized Phase II/III Trial of Prophylactic Cranial Irradiation With or Without Hippocampal Avoidance for Small Cell Lung Cancer
Brief Title: Whole-Brain Radiation Therapy With or Without Hippocampal Avoidance in Limited Stage or Extensive Stage Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRG-CC003; NCI-2015-01548 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-CC003 (Other: NRG Oncology); NRG-CC003 (Other: DCP); UG1CA189867 (NIH)
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Results first posted 2024-06-27 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Extensive Stage Small Cell Lung Carcinoma; Limited Stage Small Cell Lung Carcinoma
MeSH Terms: interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI using 3DCRT (Active Comparator): Prophylactic cranial irradiation (PCI) using three-dimensional conformal radiation therapy (3DCRT) for 2 weeks, 5 fractions/week.
  Interventions: Radiation: Three-Dimensional Conformal Radiation Therapy
- PCI with HA using IMRT (Experimental): PCI with hippocampal avoidance (HA) using intensity-modulated radiation therapy (IMRT) for 2 weeks, 5 fractions/week.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Three-Dimensional Conformal Radiation Therapy — daily fractions
  Other Names: 3-dimensional conformal radiation therapy; 3-dimensional radiation therapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; 3DCRT
  Arms: PCI using 3DCRT
Radiation: Intensity-Modulated Radiation Therapy — daily fractions
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: PCI with HA using IMRT

SUMMARY:
This randomized phase II/III trial studies how well whole-brain radiation therapy works and compares it with or without hippocampal avoidance in treating patients with small cell lung cancer that is found in one lung, the tissues between the lungs, and nearby lymph nodes only (limited stage) or has spread outside of the lung in which it began or to other parts of the body (extensive stage). Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. The hippocampus is part of the brain that is important for memory. Avoiding the hippocampus during whole-brain radiation could decrease the chance of side effects on memory and thinking. It is not yet known whether giving whole-brain radiation therapy is more effective with or without hippocampal avoidance in treating patients with small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether the 12-month intracranial relapse rate following hippocampal avoidance (HA)-prophylactic cranial irradiation (PCI) is non-inferior compared to the rate following PCI for patients with small cell lung cancer (SCLC). (Randomized Phase II Component [Non-Inferiority]) II. Determine whether HA-PCI reduces the likelihood of 6-month deterioration from baseline in Hopkins Verbal Learning Test (HVLT)-Revised (R) delayed recall compared to PCI for patients with SCLC. (Phase III Component [Efficacy])

SECONDARY OBJECTIVES:

I. Compare time to cognitive failure, as measured by a battery of tests (HVLT-R, Controlled Oral Word Association (COWA) test, and Trail Making Test (TMT) parts A and B), after PCI versus HA-PCI in SCLC.

II. Compare time to cognitive failure as separately measured by each test (HVLT-R for Total Recall and Delayed Recognition, COWA test, and TMT parts A and B), after PCI versus HA-PCI for SCLC.

III. Compare patient-reported cognitive functioning and other quality of life domains (assessed by the European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire (QLQ)-Core [C]30 and BN20) between PCI versus HA-PCI for patients with SCLC.

IV. Compare overall survival after PCI versus HA-PCI for patients with SCLC.

V. Compare 12-month intracranial relapse rate (at completion of phase III) and time to intracranial relapse after PCI versus HA-PCI for patients with SCLC.

VI. Evaluate adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) criteria.

VII. Correlate changes in health-related quality of life (HRQOL) domains with changes in cognitive testing outcomes following PCI versus HA-PCI for patients with SCLC.

VIII. Assess cost-effectiveness of HA-PCI (intensity modulated radiation therapy [IMRT]) and PCI (3-dimensional conformal radiation therapy [3DCRT]) using the EuroQual (EQ)-5-Dimensions (5D)-5L.

IX. Correlate miRNA signatures with cognitive failure in SCLC patients who received PCI and HA-PCI.

X. Evaluate Apolipoprotein E (APOE) genotyping as potential predictor of neurocognitive decline, hippocampal atrophy after brain irradiation and/or differential benefit from hippocampal avoidance.

XI. Evaluate baseline MR imaging biomarkers of white matter injury and hippocampal volumetry as potential predictors of cognitive decline and differential benefit from HA-PCI as compared to PCI.

TERTIARY OBJECTIVES:

I. Collect serum, whole blood, and urine for future translational research analyses.

II. Evaluate baseline magnetic resonance (MR) imaging biomarkers of white matter injury and hippocampal volumetry as potential predictors of cognitive decline and differential benefit from HA-PCI as compared to PCI.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo PCI using 3DCRT daily for 2 weeks.

ARM II: Patients undergo PCI with HA using IMRT daily for 2 weeks.

After completion of study treatment, patients are followed every 3 months for 1 year, then every 6 months until 3 years and then annually until death.

ELIGIBILITY:
Inclusion Criteria [prior to Step 1 registration]:

* Histologic proof or unequivocal cytologic proof (fine needle aspiration, biopsy or two positive sputa) of SCLC within 250 days prior to Step 1 registration

  * High-grade neuroendocrine carcinoma or combined SCLC and NSCLC is permitted.
* Patients must have received chemotherapy and be registered to Step 1 registration no earlier than 7 days and no later than 56 days after completing chemotherapy. Note:

  * Post-chemotherapy restaging imaging must be completed no more than 56 days prior to Step 1 registration.
  * For patients with extensive-stage small cell lung cancer who are being considered for consolidative thoracic radiotherapy after chemotherapy, concomitant administration of consolidative thoracic radiotherapy and protocol-specified prophylactic cranial irradiation with or without hippocampal avoidance is permitted.
* Patients must have a gadolinium contrast-enhanced three-dimensional (3D), spoiled gradient (SPGR), magnetization-prepared rapid gradient echo (MP-RAGE), or turbo field echo (TFE) MRI scan. To yield acceptable image quality, the gadolinium contrast-enhanced three-dimensional SPGR, MP-RAGE or TFE axial MRI scan must use the smallest possible axial slice thickness not exceeding 1.5 mm.

  * This MRI must be obtained within 56 days prior to Step 1 registration. Note: The MRI study is mandatory irrespective of randomization to the experimental or control arm of this study.
* Prior to chemotherapy +/- thoracic radiotherapy, patients must be defined as limited-stage or extensive-stage SCLC after clinical staging evaluation involving the following:

  1. History/physical examination;
  2. CT of the chest and abdomen with contrast (does not have to be done if the patient has had a positron emission tomography (PET) / CT scan prior to initiating chemotherapy or thoracic radiotherapy);
  3. MRI of the brain with contrast or diagnostic head CT with contrast;
  4. For patients without evidence of extensive-stage SCLC on chest and abdomen CT and brain MRI or head CT, a PET/CT or bone scan is required to confirm limited-stage SCLC.
* After chemotherapy, patients must be restaged prior to Step 1 registration using the same diagnostic work-up as required pre-chemotherapy. Repeat PET/CT or bone scan is not required. Patients must have:

  * History/physical examination within 30 days of Step 1 registration;
  * No CNS metastases (Repeat MRI required) within 56 days prior to Step 1 registration;
  * No progression in any site;
  * Radiographic partial or complete response to chemotherapy in at least one disease site within 56 days prior to Step 1 registration.

    1. If PET/CT was obtained prior to chemotherapy, either a repeat PET/CT or CT of the chest and abdomen with contrast can be obtained for response assessment.
    2. Patients who underwent resection for limited-stage SCLC prior to chemotherapy and have no radiographically evident disease for response assessment remain eligible if post-chemotherapy imaging demonstrates no progression.
* Zubrod performance status 0-2 within 30 days prior to Step 1 registration.
* Women of childbearing potential must have a negative qualitative serum pregnancy test =< 14 days prior to Step 1 registration.
* Patients who are primary English or French speakers are eligible
* Patients must sign a study-specific informed consent prior to study entry

Inclusion Criteria [prior to Step 2 registration]:

* The following baseline neurocognitive assessments must be completed and uploaded within 10 calendar days after or at the time of Step 1 registration: HVLT-R (recall, delayed recall, and recognition), TMT (Parts A and B), and COWA. The neurocognitive assessments will be uploaded into the NRG Oncology Rave System for evaluation by Neurocognitive Co-Chair. Once the upload is complete, within 3 business days, a notification email will be sent to the site to proceed to Step 2 registration. At minimum, the HVLT-R delayed recall must be able to be scored (i.e. completed without error) in order to be eligible.
* Patients must have a baseline raw score greater than 2 on the HVLT-R delayed recall as determined by central assessment by the Neurocognitive Co-Chair.

Exclusion Criteria:

* Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields
* Radiographic evidence of central nervous system (CNS) metastases
* Radiographic evidence of hydrocephalus or other architectural distortion of the ventricular system, including placement of external ventricular drain or ventriculoperitoneal shunt
* Planned concurrent chemotherapy during PCI

  * Concurrent atezolizumab permitted
* Concomitant invasive malignancy or invasive malignancy within the past five years other than non-melanomatous skin cancer; history of in situ carcinoma (e.g. ductal carcinoma in situ of breast, in situ carcinoma of the cervix, vulva or larynx) is permitted
* Contraindication to MR imaging, such as implanted metal devices or foreign bodies or severe claustrophobia
* Severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Uncontrolled, clinically significant cardiac arrhythmias
  * HIV positive with CD4 count < 200 cells/microliter;

    1. Note: Patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 30 days prior to Step 1 registration.
    2. Note: HIV testing is not required for eligibility for this protocol.
* Pregnant or lactating women or women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2027-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Vinai Gondi, Principal Investigator — NRG Oncology
Locations (285):
- United States (272):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Marin General Hospital, Greenbrae, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford HealthCare - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Yale University, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Ascension Saint Vincent Anderson, Anderson, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic Radiation Therapy-Northfield, Northfield, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health Imbert Cancer Center, Bay Shore, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Lenox Hill Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Atrium Health Cleveland/LCI-Cleveland, Shelby, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Crozer-Keystone Regional Cancer Center at Broomall, Broomall, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Crozer Regional Cancer Center at Brinton Lake, Glen Mills, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Lancaster Radiation Therapy Center, Lancaster, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Blount Memorial Hospital, Maryville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Ogden Regional Medical Center, Ogden, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (13):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Gondi V, Pugh SL, Mehta MP, Wefel JS, Tome WA, Sun AY, Grecula J, Redmond KJ, Fogh S, Gaspar L, Konski A, Bovi J, Robinson CG, Corn B, Videtic GM, Lok BH, Yoon HA, Heinzerling JH, DeNittis AS, McGarry RC, Devisetty K, Kundapur V, Wu AJ, McCarron EC, Thibault I, Simon EL, Baschnagel AM, Narayan S, Pollock J, Paulus R, Kachnic LA; NRG Oncology. Hippocampal Avoidance During Prophylactic Cranial Irradiation for Patients With Small Cell Lung Cancer: Randomized Phase II/III Trial NRG-CC003. J Clin Oncol. 2025 Nov 10;43(32):3516-3525. doi: 10.1200/JCO-25-00221. Epub 2025 Aug 11. PMID 40789106
- [Derived] Ishibashi A, Kurosaki H, Miura K, Utsumi N, Sakurai H. Influence of Modulation Factor on Treatment Plan Quality and Irradiation Time in Hippocampus-Sparing Whole-Brain Radiotherapy Using Tomotherapy. Technol Cancer Res Treat. 2021 Jan-Dec;20:15330338211045497. doi: 10.1177/15330338211045497. PMID 34632876

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were screened in order to determine whether their neurocognitive functioning was healthy enough to participate. This was defined as a score of 2 or higher on the Delayed Recall subscale of the Hopkins Verbal Learning Test (HVLT). HVLT testing was done after initial enrollment, but prior to randomization. Of 418 participants screened, 393 were randomized.
Period: Overall Study
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Started | 196 | 197
Phase II Analysis (These participants are included in the phase III analysis.) | 89 | 87
Adverse Event Population (Received radiation therapy.) | 191 | 189
Completed | 196 | 197
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT | Total
Number analyzed (Participants) | 196 | 197 | 393
Age, Continuous [Median (Full Range); unit: years] | 64 [34 to 84] | 65 [42 to 85] | 64 [34 to 85]
Age, Customized [Count of Participants; unit: Participants]
  Age (years): ≤ 49 | 12 | 8 | 20
  Age (years): 50-59 | 49 | 37 | 86
  Age (years): 60-69 | 75 | 102 | 177
  Age (years): ≥ 70 | 60 | 50 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 114 | 241
  Male | 69 | 83 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 185 | 190 | 375
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 10 | 25
  White | 175 | 180 | 355
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 5 | 8
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 79 | 83 | 162
    1 | 100 | 105 | 205
    2 | 17 | 9 | 26
Planned concurrent memantine use [Count of Participants; unit: Participants]
  No | 96 | 102 | 198
  Yes | 100 | 95 | 195
Extent of disease [Count of Participants; unit: Participants] — A definition of these terms was not provided in the protocol and the study sites could interpret the terms differently. LD generally refers to disease confined to the hemithorax of origin, the mediastinum, or the supraclavicular nodes and which can be encompassed within a tolerable radiation therapy port. There is no general agreement on pleural effusion, massive pulmonary tumor, and contralateral supraclavicular nodes. ED generally refers to disease that has spread beyond the supraclavicular areas and is too widespread to be considered LD. Distant metastases always indicate ED.
  Participants
    Limited stage disease (LD) | 142 | 133 | 275
    Extensive stage disease (ED) | 54 | 64 | 118
Education level [Count of Participants; unit: Participants]
  Grade school | 9 | 2 | 11
  More than grade school and did not graduate high school | 30 | 17 | 47
  High school graduate or GED | 73 | 79 | 152
  Some college or associate's degree | 46 | 64 | 110
  Bachelor's degree | 23 | 23 | 46
  Advanced degree | 14 | 9 | 23
  Unknown | 1 | 3 | 4
Smoking status (self-reported) [Count of Participants; unit: Participants]
  Never smoked | 5 | 5 | 10
  Former smoker | 62 | 61 | 123
  Current smoker | 106 | 110 | 216
  Unknown | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Deterioration in HVLT-R Delayed Recall Score at Six Months (Phase III)
Description: The HVLT-R delayed recall test assesses verbal learning and memory. The test involves memorizing a list of 12 nouns for 3 consecutive trials to recall after a 20-minute delay. The score is the sum of the number of words correctly recalled and ranges from 0 to 36, with a higher score indicating better functioning. Deterioration is defined a decrease from baseline of at least 3 points.
Time Frame: Baseline and six months
Population: Randomized patients with score at baseline and 6 months
Measure: Count of Participants; unit: Participants
Groups:
- PCI Using 3DCRT (Arm 1): Prophylactic cranial irradiation (PCI) using three-dimensional conformal radiation therapy (3DCRT) for 2 weeks, 5 fractions/week.
- PCI With HA Using IMRT (Arm 1): PCI with hippocampal avoidance (HA) using intensity-modulated radiation therapy (IMRT) for 2 weeks, 5 fractions/week.
Arm/Group | PCI Using 3DCRT (Arm 1) | PCI With HA Using IMRT (Arm 1)
Number analyzed (Participants) | 110 | 106
Participants | 33 | 27
Statistical Analysis 1: Comparison: PCI Using 3DCRT (Arm 1) vs PCI With HA Using IMRT (Arm 1); Proportion of participants with deterioration in HVLT-R delayed recall score at six months: Null hypothesis = No difference between the arms; Alternative hypothesis = Arm 2 will have less deterioration than Arm 1. Ninety-eight evaluable participants per arm at six months provides 80% statistical power to detect a 14.5% absolute difference between the arms in proportion of participants with deterioration at six months using a one-sided Fisher's exact test; Test type: Superiority; p = 0.28, Fisher Exact; one-sided significance level = 0.05

2. Primary Outcome: Number of Participants With Intracranial Relapse at 12 Months (Phase II)
Description: Intracranial relapse, defined as the development of a new brain metastasis as documented on brain MRI with contrast or head CT with contrast.
Time Frame: From baseline to 12 months
Population: Phase II randomized participants on study for at least one year.
Measure: Count of Participants; unit: Participants
Groups:
- PCI With HA Using IMRT (Arm 2): PCI with hippocampal avoidance (HA) using intensity-modulated radiation therapy (IMRT) for 2 weeks, 5 fractions/week.
Arm/Group | PCI Using 3DCRT (Arm 1) | PCI With HA Using IMRT (Arm 2)
Number analyzed (Participants) | 86 | 85
Participants | 16 | 12
Statistical Analysis 1: Comparison: PCI Using 3DCRT (Arm 1) vs PCI With HA Using IMRT (Arm 2); Test type: Non-Inferiority — Null hypothesis: Proportion of participants with relapse on Arm 2 - Arm 1 > 20%; Alternative hypothesis: Proportion of participants with relapse on Arm 2 - Arm 1 = 4.5%. Using a non-inferiority margin of 20% and an assumed difference in proportions of 4.5% under the alternative, a 2-sample test of difference in proportions with a 1-sided alpha of 0.1 requires 164 patients to achieve 85% statistical power. (Statistically significant p-value indicates non-inferiority.); p = 0.0030, Test of binomial proportions

3. Secondary Outcome: Percentage of Participants With Neurocognitive Failure (Phase III)
Description: Neurocognitive failure is defined as the first instance of neurocognitive decline in any of six assessments, as determined my reliable change index: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Recall, HVLT-R Delayed Recall, HVLT-R Delayed Recognition, Trail Making Test (TMT) part A, TMT part B, and Controlled Oral Word Association (COWA). Failure time is defined as time from randomization to failure, death (competing event), or last follow-up (censored). Neurocognitive failure rates are estimated using the cumulative incidence method. The distributions of failure times are compared, which is reported in the statistical analysis results. Six-month rates are reported here. Analysis occurred after all patients had been on study for at least six months.
Time Frame: Randomization to date of failure, death, or last known follow-up whichever occurred first. Maximum follow-up at time of analysis was 7.2 years.
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 196 | 197
percentage of participants | 57.0 [49.6 to 63.8] | 52.7 [45.3 to 59.5]
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.0598, Gray's test

4. Secondary Outcome: Number of Participants With Deterioration in HVLT-R Total Recall Score (Phase III)
Description: The HVLT-R Total Recall score assesses verbal learning and memory. The test involves memorizing a list of 12 nouns for 3 consecutive trials. Raw score is the sum of the number of targets correctly recalled, ranging from 0 to 36. Higher score indicates better functioning. Deterioration is defined a decrease from baseline of at least 5 points.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 146 | 145
Participants
  3 months: number analyzed (Participants) | 133 | 127
  3 months | 47 | 47
  6 months: number analyzed (Participants) | 110 | 106
  6 months | 33 | 35
  12 months: number analyzed (Participants) | 80 | 72
  12 months | 20 | 17
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.78, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.63, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.84, Chi-squared

5. Secondary Outcome: Number of Participants With Deterioration in HVLT-R Total Recall Score (Phase III)
Description: he HVLT-R Total Recall score assesses verbal learning and memory. The test involves memorizing a list of 12 nouns for 3 consecutive trials. Raw score is the sum of the number of targets correctly recalled, ranging from 0 to 36. Higher score indicates better functioning. Deterioration is defined a decrease from baseline of at least 5 points.
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Number of Participants With Deterioration in HVLT-R Delayed Recall Score (Phase III)
Description: The HVLT-R Delayed Recall test assesses verbal learning and memory. After memorizing a list of 12 nouns for 3 consecutive trials, this test requires recalling the 12 targets after a 20-minute delay. Raw scores are sum of the number of targets correctly recalled. The score ranges from 0 to 12. A higher score indicates better functioning. Deterioration is defined a decrease from baseline of at least 3 points. Six-month results are reported as the primary endpoint.
Time Frame: Baseline, 3, 12 months.
Population: Randomized patients with HVLT-R Delayed Recall score at baseline and: 3 or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 146 | 145
Participants
  3 months: number analyzed (Participants) | 133 | 127
  3 months | 40 | 34
  12 months: number analyzed (Participants) | 80 | 72
  12 months | 23 | 19
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.56, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.75, Chi-squared

7. Secondary Outcome: Number of Participants With Deterioration in HVLT-R Delayed Recall Score (Phase III)
Description: The HVLT-R Delayed Recall test assesses verbal learning and memory. After memorizing a list of 12 nouns for 3 consecutive trials, this test requires recalling the 12 targets after a 20-minute delay. Raw scores are sum of the number of targets correctly recalled. The score ranges from 0 to 12. A higher score indicates better functioning. Deterioration is defined a decrease from baseline of at least 3 points.
Time Frame: Baseline, 18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Number of Participants With Deterioration in HVLT-R Delayed Recognition Score (Phase III)
Description: The HVLT-R Delayed Recognition assesses verbal learning and memory. After memorizing a list of 12 nouns for 3 consecutive trials and recalling the 12 targets after a 20-minute delay, the test involves then identifying the 12 targets from a list of semantically related or unrelated items (delayed recognition). Raw scores are the sum of targets incorrectly identified subtracted from the sum of the number of targets correctly identified. The score ranges from -12 to 12 for recognition. A higher score indicates better functioning. Deterioration is defined a decrease from baseline of at least 2 points.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and: 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 146 | 145
Participants
  3 months: number analyzed (Participants) | 133 | 127
  3 months | 49 | 45
  6 months: number analyzed (Participants) | 110 | 106
  6 months | 11 | 11
  12 months: number analyzed (Participants) | 80 | 72
  12 months | 19 | 22
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.81, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.93, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.35, Chi-squared

9. Secondary Outcome: Number of Participants With Deterioration in HVLT-R Delayed Recognition Score (Phase III)
Description: as for outcome 8
Time Frame: Baseline, 18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Number of Participants With Deterioration in Trail Making Test (TMT) Part A (Phase III)
Description: The TMT is a neuropsychological test of visual attention and task switching that can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. There are two parts to the test: in the first (Part A, reported here), the targets are all numbers (1, 2, 3, etc.) and the test taker needs to connect them in sequential order. The score is the amount of time, in seconds, that it takes the patient to complete the maze. The range for Part A is 0 to 180 (3 minutes). Lower scores indicate better functioning. Deterioration is defined an increase from baseline of at least 12 seconds.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with TMT Part A at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 144 | 144
Participants
  3 months: number analyzed (Participants) | 131 | 126
  3 months | 27 | 30
  6 months: number analyzed (Participants) | 104 | 105
  6 months | 21 | 26
  12 months: number analyzed (Participants) | 78 | 70
  12 months | 22 | 14
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.54, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.43, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.25, Chi-squared

11. Secondary Outcome: Number of Participants With Deterioration in Trail Making Test (TMT) Part A (Phase III)
Description: as for outcome 10
Time Frame: Baseline, 18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: Number of Participants With Deterioration in TMT Part B Score (Phase III)
Description: The TMT is a neuropsychological test of visual attention and task switching that can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. There are two parts to the test: in the second part (Part B, reported here), the subject alternates between numbers and letters (1, A, 2, B, etc.). The score is the amount of time, in seconds, that it takes the patient to complete the maze. The score range for Part B is 0 to 300 (5 minutes). Lower scores indicate better functioning. Deterioration is defined an increase from baseline of at least 26 seconds.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 142 | 143
Participants
  3 months: number analyzed (Participants) | 127 | 120
  3 months | 43 | 38
  6 months: number analyzed (Participants) | 103 | 104
  6 months | 26 | 38
  12 months: number analyzed (Participants) | 76 | 69
  12 months | 22 | 19
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.71, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.079, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.85, Chi-squared

13. Secondary Outcome: Number of Participants With Deterioration in TMT Part B Score (Phase III)
Description: The TMT is a neuropsychological test of visual attention and task switching that can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. There are two parts to the test: in the second part (Part B, reported here), the subject alternates between numbers and letters (1, A, 2, B, etc.). The score is the amount of time, in seconds, that it takes the patient to complete the maze. The score range for Part B is 0 to 300 (5 minutes). Lower scores indicate better functioning. Deterioration is defined an increase from baseline of at least 26 seconds.
  If reporting a score on a scale, please include the unabbreviated scale title, the minimum and maximum values, and whether higher scores mean a better or worse outcome.
Time Frame: Baseline, 18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

14. Secondary Outcome: Number of Participants With Deterioration in Controlled Oral Word Association (COWA) Score (Phase III)
Description: The COWA is a verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with some designated letter. Patients are given 1 minute to name as many words as possible beginning with the designated letter. The procedure is then repeated for the remaining two letters. Two alternate forms of the COWA are employed to minimize practice effects. The score is the sum of the correct responses with a range of 0 to infinity. A higher score indicates better functioning. Deterioration is defined an increase from baseline of at least 12 words.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 145 | 145
Participants
  3 months: number analyzed (Participants) | 132 | 129
  3 months | 13 | 24
  6 months: number analyzed (Participants) | 109 | 108
  6 months | 3 | 12
  12 months: number analyzed (Participants) | 81 | 73
  12 months | 7 | 14
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.043, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.017, Fisher Exact
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12-month; Test type: Superiority; p = 0.057, Chi-squared

15. Secondary Outcome: Number of Participants With Deterioration in Controlled Oral Word Association (COWA) Score (Phase III)
Description: as for outcome 14
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

16. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported (Phase III)
Description: Common Terminology Criteria for Adverse Events (version 5) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From start of treatment to last known follow-up . Maximum follow-up time was 7.2 years.
Population: Randomized participants who received radiation therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 191 | 189
Participants
  Grade 1 | 27 | 30
  Grade 2 | 78 | 75
  Grade 3 | 47 | 47
  Grade 4 | 12 | 8
  Grade 5 | 1 | 3

17. Secondary Outcome: Number of Participants With Deterioration in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (QLQ-C30) Global Health Status (Phase III)
Description: The QLQ-C30 is a 30-item self-report questionnaire used to assess the health-related quality of life (QOL) of cancer patients participating in international clinical trials. Global Health Status is considered a measure of overall quality of life and is calculated from two questions whose raw scores are averaged and then transformed to a range of 0 (worst) to 100 (best). Deterioration is defined a reduction of 10% from baseline.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 146 | 137
Participants
  3 months: number analyzed (Participants) | 129 | 123
  3 months | 57 | 67
  6 months: number analyzed (Participants) | 115 | 107
  6 months | 39 | 43
  12 months: number analyzed (Participants) | 84 | 77
  12 months | 22 | 26
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.10, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.33, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.29, Chi-squared

18. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Global Health Status (Phase III)
Description: as for outcome 17
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

19. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Physical Functioning Score (Phase III)
Description: The EORTC QLQ-C30 is a 30-item self-report questionnaire used to assess the health-related quality of life of cancer patients participating in international clinical trials. A functional scale raw score is transformed to a range of 0 (worst) to 100 (best) in which a high score represents a healthy level of functioning. Deterioration is defined a reduction of 10% from baseline.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 147 | 137
Participants
  3 months: number analyzed (Participants) | 129 | 122
  3 months | 39 | 60
  6 months: number analyzed (Participants) | 116 | 107
  6 months | 30 | 46
  12 months: number analyzed (Participants) | 85 | 77
  12 months | 25 | 28
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.0021, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.0070, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.35, Chi-squared

20. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Physical Functioning Score (Phase III)
Description: as for outcome 19
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

21. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Role Functioning Score (Phase III)
Description: The EORTC QLQ-C30 is a 30-item self-report questionnaire used to assess the health-related quality of life (QOL) of cancer patients participating in international clinical trials. A functional scale raw score is transformed to a range of 0 (worst) to 100 (best) in which a high score represents a healthy level of functioning. Deterioration is defined a reduction of 10% from baseline.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 147 | 137
Participants
  3 months: number analyzed (Participants) | 127 | 121
  3 months | 54 | 56
  6 months: number analyzed (Participants) | 113 | 107
  6 months | 30 | 41
  12 months: number analyzed (Participants) | 83 | 77
  12 months | 20 | 24
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.55, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.062, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.32, Chi-squared

22. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Role Functioning Score (Phase III)
Description: as for outcome 21
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

23. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Emotional Functioning Score (Phase III)
Description: as for outcome 19
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 147 | 137
Participants
  3 months: number analyzed (Participants) | 129 | 123
  3 months | 46 | 41
  6 months: number analyzed (Participants) | 115 | 107
  6 months | 31 | 33
  12 months: number analyzed (Participants) | 85 | 77
  12 months | 19 | 19
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.70, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.52, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.73, Chi-squared

24. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Emotional Functioning Score (Phase III)
Description: as for outcome 19
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

25. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Social Functioning Score (Phase III)
Description: as for outcome 21
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 147 | 137
Participants
  3 months: number analyzed (Participants) | 124 | 121
  3 months | 39 | 46
  6 months: number analyzed (Participants) | 110 | 104
  6 months | 21 | 30
  12 months: number analyzed (Participants) | 83 | 75
  12 months | 17 | 13
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.28, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.094, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.61, Chi-squared

26. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Social Functioning Score (Phase III)
Description: as for outcome 21
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

27. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Cognitive Functioning Score (Phase III)
Description: as for outcome 21
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT (Arm 1) | PCI With HA Using IMRT (Arm 2)
Number analyzed (Participants) | 147 | 137
Participants
  3 months: number analyzed (Participants) | 127 | 122
  3 months | 58 | 45
  6 months: number analyzed (Participants) | 114 | 106
  6 months | 41 | 55
  12 months: number analyzed (Participants) | 84 | 76
  12 months | 37 | 30
Statistical Analysis 1: Comparison: PCI Using 3DCRT (Arm 1) vs PCI With HA Using IMRT (Arm 2); 3 months; Test type: Superiority; p = 0.16, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT (Arm 1) vs PCI With HA Using IMRT (Arm 2); 6 months. Assuming 50% of patients experience deterioration at 6 months, based on a prior study (RTOG-0212), a sample size of 198 participants per arm provides 94% power to detect a 50% relative reduction (50% on Arm 1 vs. 25% on Arm 2) in decline at 6 months using Fisher's exact test with a two-sided alpha=0.05; Test type: Superiority; p = 0.017, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT (Arm 1) vs PCI With HA Using IMRT (Arm 2); 12-month; Test type: Superiority; p = 0.56, Chi-squared

28. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-C30 Cognitive Functioning Score (Phase III)
Description: as for outcome 21
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

29. Secondary Outcome: Number of Participants With Deterioration in EORTC Quality of Life Questionnaire BN-20 (QLQ-BN20) Motor Dysfunction Score (Phase III)
Description: The EORTC QLQ-BN20 is a 20-item self-report questionnaire supplement to the QLQ-C30 for patients used to assess the health-related quality of life of brain cancer patients. A symptom scale raw score is transformed to a range of 0 (best) to 100 (worst) in which a high score represents a high level of symptomatology/problems. For patients with a baseline score of 0, a follow-up score of ≥ 10 is considered as a deterioration. Otherwise, a 10% increase is considered as a deterioration.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 149 | 140
Participants
  3 months: number analyzed (Participants) | 132 | 125
  3 months | 57 | 60
  6 months: number analyzed (Participants) | 115 | 107
  6 months | 49 | 51
  12 months: number analyzed (Participants) | 86 | 79
  12 months | 37 | 41
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.44, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.45, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.25, Chi-squared

30. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-BN20 Motor Dysfunction Score (Phase III)
Description: as for outcome 29
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

31. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-BN20 Communication Deficit Score (Phase III)
Description: The QLQ-BN20 is a 20-item self-report questionnaire supplement to the QLQ-C30 for patients used to assess the health-related quality of life of brain cancer patients. A symptom scale raw score is transformed to a range of 0 (best) to 100 (worst) in which a high score represents a high level of symptomatology/problems. For patients with a baseline score of 0, a follow-up score of ≥ 10 is considered as a deterioration. Otherwise, a 10% increase is considered as a deterioration.
Time Frame: Baseline, 3, 6, 12 months.
Population: Randomized patients with score at baseline and 3, 6, or 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 149 | 140
Participants
  3 months: number analyzed (Participants) | 132 | 124
  3 months | 50 | 40
  6 months: number analyzed (Participants) | 115 | 107
  6 months | 45 | 42
  12 months: number analyzed (Participants) | 86 | 79
  12 months | 31 | 28
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 3 months; Test type: Superiority; p = 0.35, Chi-squared
Statistical Analysis 2: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 6 months; Test type: Superiority; p = 0.99, Chi-squared
Statistical Analysis 3: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; 12 months; Test type: Superiority; p = 0.94, Chi-squared

32. Secondary Outcome: Number of Participants With Deterioration in EORTC QLQ-BN20 Communication Deficit Score (Phase III)
Description: as for outcome 31
Time Frame: Baseline,18, 24 months.
Reporting Status: Not Posted, anticipated posting 2025-12

33. Secondary Outcome: Correlation of Quality of Life and Neurocognitive Function (NCF) Measures at 6 Months
Description: The Pearson correlation coefficient was calculated for EORTC QLQ-C30 (physical, role, emotional, cognitive, and social functioning domains and global health status) and QLQ-BN20 (motor dysfunction and communication deficit) versus the standardized neurocognitive function (HVLT-R total recall, HVLT-R delayed recall, HVLT-R delayed recognition, COWA, TMT parts A and B) and the Clinical Trial Battery Composite (CTB Comp) score (mean of the z-scores for the six NCF scores) for all patients, treatment arms combined. The Pearson correlation coefficient is computed for each pair of measurements, resulting in 48 correlation coefficients. Possible values range from -1 (negatively correlated) to 1(positively correlated), with 0 indicating no correlation. A correlation with a value in range -0.35 to 0.35 is considered weak and is indicated by "0" in the table. Because of the large number of comparisons, only individual correlation coefficients outside that range are listed here.
Time Frame: 6 months
Population: Randomized participants with values at 6 months. The protocol specifies that the treatment arms are combined into a single group for this outcome measure.
Measure: Number; unit: correlation coefficient
Groups:
- Participants Combined From Both Arms: Prophylactic cranial irradiation (PCI) using three-dimensional conformal radiation therapy (3DCRT) for 2 weeks, 5 fractions/week.
  PCI with hippocampal avoidance (HA) using intensity-modulated radiation therapy (IMRT) for 2 weeks, 5 fractions/week.
Arm/Group | Participants Combined From Both Arms
Number analyzed (Participants) | 212
correlation coefficient
  EORTC QLQ-C30 Physical functioning vs. NCF CTB Comp Score: number analyzed (Participants) | 207
  EORTC QLQ-C30 Physical functioning vs. NCF CTB Comp Score | 0.3619
  All others | 0

34. Secondary Outcome: Incremental Cost-per Quality-adjusted Life Year (QALY) (Cost-effectiveness as Measured by the EQ-5D (Phase III)
Description: The incremental cost per quality-adjusted life year (QALY) ratio will be calculated as total cost of the PCI with HA using IMRT arm (Arm 2) minus total cost of the PCI using 3DCRT arm (Arm 1), divided by the quality adjusted survival of the Arm 1 patients minus the quality adjusted survival of Arm 2 patients.
Time Frame: Baseline to two years
Reporting Status: Not Posted, anticipated posting 2025-12

35. Secondary Outcome: Overall Survival (Phase III)
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated by the Kaplan-Meier method. Analysis occurred after all patients had been on study for at least 8 months.
Time Frame: From the date of randomization to the date of death or last follow-up. Maximum follow-up time at time of analysis was 7.2 years.
Population: Randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 196 | 197
months | 24.9 [17.8 to 36.4] | 20.7 [17.0 to 34.7]
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.79, Log Rank — Two-side significance level = 0.05

36. Secondary Outcome: Intracranial Relapse Rate (Phase III)
Description: Intracranial relapse is defined as the development of a new brain metastasis as documented on brain MRI with contrast or head CT with contrast. Time to intracranial relapse is defined as time from randomization to the date of first intracranial relapse, last known follow-up (censored), or death without intracranial relapse (competing risk), whichever occurred first. Intracranial relapse rates are estimated using the cumulative incidence method. The distributions of intracranial relapse times are compared between the arms, which is reported in the statistical analysis results. One-year rates are provided here. Analysis occurred at time of the phase III primary analysis.
Time Frame: From date of randomization to date of intracranial relapse, death, or last known follow-up, whichever occurred first. Maximum follow-up at time of analysis was 7.2 years.
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
Number analyzed (Participants) | 196 | 197
percentage of participants | 15.9 [11.0 to 21.6] | 15.7 [10.9 to 21.4]
Statistical Analysis 1: Comparison: PCI Using 3DCRT vs PCI With HA Using IMRT; Test type: Superiority; p = 0.93, Gray's test

37. Secondary Outcome: White Matter Injury and Hippocampal Volume on Neurocognitive Function (Phase III)
Description: Pearson correlation coefficients will be used to assess the effect of hippocampal volume and FLAIR volume change on baseline neurocognitive function, as measured by the HVLT-R, COWA, and TMT, separately for each arm.
Time Frame: Baseline to 6 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Baseline to last known follow-up or death. Maximum follow-up time was 7.2 years.
Description: All-cause mortality was assessed in randomized participants. Adverse events were assessed in randomized participants who started radiation therapy.
Arm/Group | PCI Using 3DCRT | PCI With HA Using IMRT
All-Cause Mortality (participants affected / at risk) | 118/196 | 112/197
Serious Adverse Events (participants affected / at risk) | 26/191 | 17/189
Other Adverse Events (participants affected / at risk) | 154/191 | 152/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PCI Using 3DCRT (N=191) | PCI With HA Using IMRT (N=189)
Anemia (Blood and lymphatic system disorders) | 0 | 4
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Endocrine disorders - Other (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 3
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Chills (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 2
Fatigue (General disorders) | 3 | 3
Fever (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 1
Serum sickness (Immune system disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 5 | 3
Otitis media (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 2
Weight loss (Investigations) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 2
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PCI Using 3DCRT (N=191) | PCI With HA Using IMRT (N=189)
Anemia (Blood and lymphatic system disorders) | 24 | 18
Hearing impaired (Ear and labyrinth disorders) | 24 | 11
Tinnitus (Ear and labyrinth disorders) | 12 | 6
Blurred vision (Eye disorders) | 21 | 16
Constipation (Gastrointestinal disorders) | 34 | 19
Diarrhea (Gastrointestinal disorders) | 16 | 17
Dry mouth (Gastrointestinal disorders) | 10 | 12
Dysphagia (Gastrointestinal disorders) | 16 | 9
Nausea (Gastrointestinal disorders) | 69 | 61
Vomiting (Gastrointestinal disorders) | 31 | 26
Fatigue (General disorders) | 116 | 103
Gait disturbance (General disorders) | 16 | 16
Pain (General disorders) | 19 | 15
Dermatitis radiation (Injury, poisoning and procedural complications) | 28 | 14
Fall (Injury, poisoning and procedural complications) | 17 | 12
Lymphocyte count decreased (Investigations) | 20 | 11
Platelet count decreased (Investigations) | 13 | 10
Weight loss (Investigations) | 26 | 26
Anorexia (Metabolism and nutrition disorders) | 38 | 39
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 18
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 20 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 7
Amnesia (Nervous system disorders) | 10 | 4
Dizziness (Nervous system disorders) | 46 | 48
Dysgeusia (Nervous system disorders) | 20 | 16
Headache (Nervous system disorders) | 74 | 73
Memory impairment (Nervous system disorders) | 41 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 14
Anxiety (Psychiatric disorders) | 15 | 11
Confusion (Psychiatric disorders) | 8 | 11
Depression (Psychiatric disorders) | 13 | 12
Insomnia (Psychiatric disorders) | 18 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 39 | 38
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 49 | 52
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 42 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 7

LIMITATIONS AND CAVEATS:
Phase II participants were included in the phase III analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02635009/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT02635009/ICF_001.pdf